CLINICAL TRIAL: NCT01550874
Title: STEP: Enhanced Physical Activity in Children and Youth With Epilepsy: Developing Evidence of Impacts on Health, Functioning, Psychological Wellbeing, and Quality of Life
Brief Title: STEP: Enhanced Physical Activity in Children and Youth With Epilepsy
Acronym: STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Academic Health Sciences Organization (Other); Ontario Brain Institute (Other); The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: REB 12-035; NCT01889901 (obsolete NCT alias)
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Epilepsy
Keywords: Physical Activity; Epilepsy; Children; Motivation
MeSH Terms: conditions — Epilepsy; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Wear the pedometer provided by study everyday with weekly charging and syncing of data.
- Experimental Group (Experimental): Wear the pedometer provided by the study everyday and also participate in phone-based physical activity behavior-change counselling for 6 months and then check sustainability without further motivational support for another 6 months.
  Interventions: Behavioral: Physical activity behavior-change counselling

INTERVENTIONS:
Behavioral: Physical activity behavior-change counselling — Participants in the experimental group will be motivated by augmented behavior modification strategies aiming to increase performance by: (i) having access to the pedometer web page that allows them to view their automatically calculated goals, and (ii) get feedback about performance toward goals.
  Arms: Experimental Group

SUMMARY:
Epilepsy is common in childhood. Children with epilepsy are at increased risk of impaired health, functioning, psychological well-being, and quality of life. There is compelling evidence that physical activity improves the medical and psychosocial aspects of health in adults with epilepsy - but there are no such studies in children. This study is to see if increased levels of physical activity can influence children's functioning, psychological well-being, and quality of life.

DETAILED DESCRIPTION:
There are many unfounded assumptions about the dangers of exercise in children with epilepsy - assumptions that may be seriously detrimental to children's health, and that we have good reason to challenge. This project explores the innovative idea that enhancing physical activity in children with epilepsy will have a positive effect on medical and psychosocial outcomes. The primary purpose of this study is to examine whether increasing physical activity levels through a six-month walking program, that includes behavioral counselling and self-monitoring of physical activity, as compared to varied un-standardized current practices, positively influences health and quality of life over one year. The secondary purposes are to (i) determine which environmental and personal facilitators and barriers to physical activity are experienced when increasing physical activity levels through a six-month walking program; (ii) determine if physical activity levels established during the six-month program will be sustained over a subsequent six-month period that includes self-monitoring of physical activity only; (iii) identify aspects of health that are amendable to change with enhanced physical activity, and explore the relationships among physical activity and impairments, functioning, psychological well-being and quality of life; and (iv) assess if there is a dose-response relationship between physical activity and a variety of health and social factors and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Has epilepsy, as confirmed by a pediatric neurologist, with at least 1 seizure in the previous 12 months
* Ambulatory
* Fluency English or French
* Intellectual functioning at or greater than grade 3 level, as judged by parents
* Access to a computer

Exclusion Criteria:

* Additional diagnoses of psychogenic seizures or autism
* Enrolled in a potentially confounding trial

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2012-04-02 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
CHEQOL-25 | Baseline, 16 week follow-up, 28 week follow-up
  Measure of quality of life
KIDSCREEN-27 | Baseline, 16 week follow-up, 28 week follow-up
  Will look at Psychological Well-Being (7items) subscale
Step Count | Baseline, 16 week follow-up, 28 week follow-up
  Will use step counts obtained from pedometer

SECONDARY OUTCOMES:
KIDSCREEN-27 | Baseline, 16 week follow-up, 28 week follow-up
  Will look at Physical Well-Being (5 items), Parents and Autonomy (7 items), Social Support and Peers (4 items) and School Environment (4 items) subscales

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel M Ronen, MD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No